CLINICAL TRIAL: NCT05704777
Title: Impact of Physical Activity as a Coadjuvant Strategy to Pharmacological Treatment for Glaucoma Management: A Randomized Clinical Trial in Primary Open-angle Glaucoma Patients (EYE-FIT)
Brief Title: Exercise Intervention in Primary Open-angle Glaucoma
Acronym: EYE-FIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Granada (Other)
Collaborators: University Hospital Virgen de las Nieves (Other); Durham University (Other); University of Szczecin (Unknown)
Responsible Party: Principal Investigator, Jesus Vera Vilchez, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PID2021-127505NA-I00; PID2021-127505NA-I00 (Other Grant/Funding Number: Ministerio de Ciencia e Innovación)
Record Dates: First submitted 2022-12-30; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Glaucoma, Open-Angle; Glaucoma
Keywords: Exercise; Multidisciplinary intervention; Eye care
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: The assessment of the outcomes will be performed by researchers blinded to the group allocation of each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise (Experimental): The intervention (endurance + resistance training) group will perform 48 training sessions (24 weeks, twice per week). In each session, they will perform the leg and arm cycling exercises during the first half of the session (15 minutes of leg cycling and 15 minutes of arm cycling) and resistance training exercises involving the lower-body (e.g., squat) and upper-body (e.g., a variety exercises performed against the resistance imposed by elastic bands) during the second half of the session.
  Interventions: Behavioral: Exercise; Other: Control
- control (No Intervention): The control group will not perform any supervised training program, and will follow standard care.

INTERVENTIONS:
Behavioral: Exercise — A 24-weeks concurrent exercise training program
  Arms: exercise
Other: Control — Usual care
  Arms: exercise

SUMMARY:
EYE-FIT is a randomized clinical trial with a two-arm parallel design aimed at assessing the impact of performing a structured and supervised physical training program on the different variables associated with glaucoma progression in pharmacologically treated primary open angle glaucoma patients. This intervention will include a supervised 24-weeks concurrent (endurance + resistance) training program comparing its influence to the standard care.

DETAILED DESCRIPTION:
There are claims that more physically active individuals are less likely to glaucoma onset and progression. However, to date, there is not a single randomized controlled clinical trial assessing the impact of performing a structured and supervised physical training program on glaucoma progression. A randomized controlled clinical trial with a two-arm parallel design will be used to determine the chronic effects of a 24-weeks concurrent (endurance + resistance) training program in comparison to a control group (no training prescribed) on the ocular function and physical fitness of primary open angle glaucoma patients. Participants will be randomly divided in one of the two groups (experimental or control [wait-list]), while ocular function and physical fitness will be assessed before and after the intervention by researchers blinded to the group allocation of each participant. In addition, primary open angle glaucoma patients will be subdivided according to their medical treatment in two groups (prostaglandin analogues and combination of prostaglandin analogue and beta-blockers). Therefore, four groups will be considered in this clinical trial. The results of the EYE-FIT clinical trial will provide novel information on the influence of exercise on different markers of glaucoma, and may help to reduce the clinical, economic and social burden of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Have an age between 50 and 70 years old
* Primary open angle glaucoma diagnosis based on objective criteria (i.e., glaucomatous optic nerve head changes and visual field defects consistent with glaucoma, after the exclusion of other possible causes).
* No have undergone any surgical intervention for glaucoma treatment
* Be medically treated with prostaglandin analogues or with a combination of prostaglandin analogue and beta-blockers

Exclusion Criteria:

* Have an scheduled surgery for the following 6 months
* Have a sufficient level of mobility to perform supervised physical exercise
* Suffer any disease that prevent the practice of physical exercise

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline glaucomatous damage in the retina at 6 months | Baseline (week 0) and after-intervention (week 25)
  Optical coherence tomography for the assessment of glaucomatous damage in the macula and optic nerve head
Change from baseline visual fields at 6 months | Baseline (week 0) and after-intervention (week 25)
  Evaluation of the visual fields with the Humphrey Field Analyzer using the Swedish Interactive Thresholding Algorithm (24-2) SITA-Standard protocol .
Changes from baseline anterior eye morphology and corneal biomechanics at 6 months | Baseline (week 0) and after-intervention (week 25)
  Assessment of the anterior chamber morphology using the Pentacam Scheimpflug camera and the biomechanics of the cornea using the Corvis ST.
Change from baseline electrophysiological activity in the retina at 6 months | Baseline (week 0) and after-intervention (week 25)
  Examination of the functional state of the retina with the photopic negative response and pattern ERG
Change from baseline intraocular pressure at 6 months | Baseline (week 0) and after-intervention (week 25)
  Assessment of intraocular pressure levels
Change from baseline ocular perfusion pressure at 6 months | Baseline (week 0) and after-intervention (week 25)
  Indirect calculation of ocular perfusion pressure by the measure of intraocular pressure and blood pressure

SECONDARY OUTCOMES:
Self-reported vision-targeted health status | Baseline (week 0) and after-intervention (week 25)
  The 25-item National Eye Institute Visual Function Questionnaire (NEI VFQ-25). Minimum value: 0 // Maximum value: 100. Higher scores mean a better outcome.
Glaucoma-specific questionnaire | Baseline (week 0) and after-intervention (week 25)
  The Glaucoma Symptom Scale (GSS). Minimum value: 0 // Maximum value: 100. Higher scores mean a better outcome.
Glaucoma-related quality of life | Baseline (week 0) and after-intervention (week 25)
  The 15-item Glaucoma Quality of Life (GQL-15). Minimum value: 0 // Maximum value: 100. Higher scores mean a worse outcome.
Health-related quality of life | Baseline (week 0) and after-intervention (week 25)
  The 36-Item Short Form Health Survey questionnaire (SF-36). Minimum value: 0 // Maximum value: 100. Higher scores mean a better outcome.
Self-rated health in mobility, self-care, usual activities, pain/discomfort and anxiety/depression | Baseline (week 0) and after-intervention (week 25)
  The EuroQol Group inventory of 5 dimensions and 3 levels (EQ-5D-3L). Minimum value: 0 // Maximum value: 1. Higher scores mean a better outcome.
Assessment of emotional (hedonic), social and psychological well-being. | Baseline (week 0) and after-intervention (week 25)
  The Mental Health Continuum-Short Form (MHC-SF). Minimum value: 0 // Maximum value: 70. Higher scores mean a better outcome.
Distress evaluation along the 3 axes of depression, anxiety and stress | Baseline (week 0) and after-intervention (week 25)
  The Depression, Anxiety and Stress Scale short form (DASS-21). Minimum value: 0 // Maximum value: 21. Higher scores mean a worse outcome.
Strength performance | Baseline (week 0) and after-intervention (week 25)
  Evaluation of the velocity recorded against submaximal loads with a linear position transducer in the squat and bench press exercises.
Endurance performance | Baseline (week 0) and after-intervention (week 25)
  An incremental loading test will be performed on a leg crank ergometer
Weight | Baseline (week 0) and after-intervention (week 25)
  Weight measured with a scale (kg).
Fat mass | Baseline (week 0) and after-intervention (week 25)
  Body composition assessment will be obtained through a segmental multi-frequency body composition analyzer. Fat mass in kg.
Lean mass | Baseline (week 0) and after-intervention (week 25)
  Body composition assessment will be obtained through a segmental multi-frequency body composition analyzer. Lean mass in kg.
Visceral adipose tissue | Baseline (week 0) and after-intervention (week 25)
  Body composition assessment will be obtained through a segmental multi-frequency body composition analyzer. Visceral adipose tissue in kg.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided